CLINICAL TRIAL: NCT03198377
Title: The Effect of Frequency Modulation in Transcutaneous Electrical Nerve Stimulation (TENS) on Habituation and Pain Threshold: a Randomized, Double Blind, Controlled Cross-over
Brief Title: The Effect of Frequency Modulation in TENS on Habituation and Pain Threshold
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Castilla-La Mancha (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: UCastillaLaMancha
Record Dates: First submitted 2017-05-23; First posted 2017-06-26 (Actual); Last update posted 2017-11-14 (Actual); Status verified 2017-07

CONDITIONS: Transcutaneous Electrical Nerve Stimulation
Keywords: Pain Threshold; Transcutaneous Electrical Nerve Stimulation; Habituation
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- TENS: Randomized frequency modulation (Experimental): TENS transcutaneous electrical stimulation over superficial radial nerve through the electrotherapy device Myomed 932. (Enraf-Nonius, Delft, Netherlands)
  Interventions: Device: TENS: Randomized frequency modulation
- TENS: Scan 6/6 of frequency modulation (Experimental): TENS transcutaneous electrical stimulation over superficial radial nerve through the electrotherapy device Myomed 932. (Enraf-Nonius, Delft, Netherlands)
  Interventions: Device: TENS: Scan 6/6 of frequency modulation
- TENS: Fixed frequency (Experimental): TENS transcutaneous electrical stimulation over superficial radial nerve through the electrotherapy device Myomed 932. (Enraf-Nonius, Delft, Netherlands)
  Interventions: Device: TENS: Fixed frequency
- TENS: Sham stimulation (Sham Comparator): Sham transcutaneous electrical stimulation over superficial radial nerve through the electrotherapy device Myomed 932. (Enraf-Nonius, Delft, Netherlands)
  Interventions: Device: Sham Stimulation

INTERVENTIONS:
Device: TENS: Randomized frequency modulation — Transcutaneous application of Conventional TENS current over the course of the superficial radial nerve in the right forearm for a 20 minutes session. The intensity of the current will increase until participants report a "strong but comfortable" sensation, just Transcutaneous application of Conventional TENS current over the course of the superficial radial nerve in the right forearm for a 20 minutes session. The intensity of the current will increase until participants report a "strong but comfortable" sensation, just below motor threshold. Currents parameters are:
  Frequency modulation: randomized pattern (from 80 to 120 Hz) Pulse width 200 microseconds
  Arms: TENS: Randomized frequency modulation
Device: TENS: Scan 6/6 of frequency modulation — Transcutaneous application of Conventional TENS current over the course of the superficial radial nerve in the right forearm for a 20 minutes session. The intensity of the current will increase until participants report a "strong but comfortable" sensation, just below motor threshold. Currents parameters are:
  Frequency modulation: Scan of frequency from 80 to 120 Hz in 6/6 mode (frequency sweep from 80 Hz to 120 Hz in 6 seconds and from 120 to 80 Hz in 6 secons) Pulse width 200 microseconds
  Arms: TENS: Scan 6/6 of frequency modulation
Device: TENS: Fixed frequency — Transcutaneous application of Conventional TENS current over the course of the superficial radial nerve in the right forearm for a 20 minutes session. The intensity of the current will increase until participants report a "strong but comfortable" sensation, just below motor threshold. Currents parameters are:
  Fixed frequency at 100 Hz Pulse width 200 microseconds
  Arms: TENS: Fixed frequency
Device: Sham Stimulation — Electrodes are placed over the course of the superficial radial nerve in the right forearm for a 20 minutes in the same manner as experimental groups, but will be applied a sham electrical stimulation increasing the current intensity of an unconnected channel.
  Arms: TENS: Sham stimulation

SUMMARY:
Purpose

The purpose of this study is to determine whether application of Transcutaneous Electrical Nerve Stimulation (TENS) is effective on habituation to electrical current whether delivered at a fixed frequency of 100 Hz or at patterned frequency. The secondary purposes are to determine the effectiveness on mechanical pressure pain and the subjective perception of the subjects regarding habituation and comfort of the different stimulations.

DETAILED DESCRIPTION:
Low frequency and low intensity TENS showed strong evidence of inefficiency while conventional high frequency TENS (around 100Hz) applied at "strong but comfortable" intensity proved strong evidence of efficacy on pressure pain. In addition, some studies have shown the importance of current intensity in the effect of TENS.

Either in clinical practice and in research, TENS intensity is usually adjusted according to the sensation of the subjects "strong but comfortable" "strong just below the motor threshold", ...). Usually throughout the TENS applications there is a phenomenon called "habituation" that involve a wide decrease of the sensation of the current applied, even though the perception the output-parameters are maintained.

In this sense, It has been seem that adjusting the intensity throughout the TENS intervention produced a greater hypoalgesic effect than when the intensity remained fixed.

On the other hand, most TENS devices offer the possibility of modulating current with the aim of preventing habituation phenomenon. The modulation of the electric current consists of changing the characteristics of the current (pulse width, pulse frequency, ...) every few seconds during the intervention. Nevertheless, the most common pattern used is the frequency modulation. However, there is a lack of evidence regarding what it is the better methods to avoid habituation during a TENS application.

ELIGIBILITY:
Inclusion Criteria:

* Participants will be volunteer healthy students of University of Castilla - La Mancha, older than 18 years.

Exclusion Criteria:

* Neuromuscular disease. Epilepsy. Trauma, surgery or pain affecting the upper limb, shoulder girdle or cervical area.

Osteosynthesis material in the upper limb. Cancer. Cardiovascular disease. Pacemaker or other implanted electrical device. Take any drug (NSAIDs, corticosteroids, antidepressants, analgesics, antiepileptics, ...) during the study and in the previous 7 days.

Presence of tattoos or other external agent introduced into the treatment or assessment area.

Pregnancy. Sensitivity disturbance in upper limb.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 39 (Actual)
Dates: Start 2017-07-03 (Actual); Primary Completion 2017-09-05 (Actual); Study Completion 2017-09-30 (Actual)

PRIMARY OUTCOMES:
Habituation to electrical stimulation | Baseline
  Due to habituation it is necessary to increase the intensity of the current throughout the session. Two measures were recorded within this variable: i) the increase in current density (mA / cm2) throughout the session (difference between its initial frequency and final frequency value of the current) and the number of times the participant requested to increase the intensity (subjects were instructed to maintain the same threshold)
Habituation to electrical stimulation | during treatment at 15 min
  Due to habituation it is necessary to increase the intensity of the current throughout the session. Two measures were recorded within this variable: i) the increase in current density (mA / cm2) throughout the session (difference between its initial frequency and final frequency value of the current) and the number of times the participant requested to increase the intensity (subjects were instructed to maintain the same threshold)
Habituation to electrical stimulation | at 10 min. post-treatment
  Due to habituation it is necessary to increase the intensity of the current throughout the session. Two measures were recorded within this variable: i) the increase in current density (mA / cm2) throughout the session (difference between its initial frequency and final frequency value of the current) and the number of times the participant requested to increase the intensity (subjects were instructed to maintain the same threshold)

SECONDARY OUTCOMES:
Mechanical pain threshold | Baseline
  The pressure pain threshold will be measured by a pressure digital algometer (Wagner Instruments, FDIX. Post Office Box 1217, Greenwich, CT 06836-1217 USA.) and will be expressed in Newton; on the back of the right hand (about 3 cm from the first interdigital foldand) . The mechanical pain threshold will be assessed 3 time in order to calculate the mean value.
Mechanical pain threshold | during treatment at 15 min.
  The pressure pain threshold will be measured by a pressure digital algometer (Wagner Instruments, FDIX. Post Office Box 1217, Greenwich, CT 06836-1217 USA.) and will be expressed in Newton; on the back of the right hand (about 3 cm from the first interdigital foldand) . The mechanical pain threshold will be assessed 3 time in order to calculate the mean value.
Mechanical pain threshold | at 10 min. post-treatment
  The pressure pain threshold will be measured by a pressure digital algometer (Wagner Instruments, FDIX. Post Office Box 1217, Greenwich, CT 06836-1217 USA.) and will be expressed in Newton; on the back of the right hand (about 3 cm from the first interdigital foldand) . The mechanical pain threshold will be assessed 3 time in order to calculate the mean value.
Perception current comfortability | at 1min. post-treatment
  Visual scale from 0 mm to 100 mm
Perception current habituation | at 1min. post-treatment
  Visual scale from 0 mm to 100 mm

CONTACTS AND LOCATIONS:
Overall Officials: Juan Avendaño-Coy, PhD, Study Director — University of Castilla-La Mancha
Locations (1):
- Juan Avendaño-Coy, Toledo, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Avendano-Coy J, Bravo-Esteban E, Ferri-Morales A, Martinez-de la Cruz R, Gomez-Soriano J. Does Frequency Modulation of Transcutaneous Electrical Nerve Stimulation Affect Habituation and Mechanical Hypoalgesia? A Randomized, Double-Blind, Sham-Controlled Crossover Trial. Phys Ther. 2019 Jul 1;99(7):924-932. doi: 10.1093/ptj/pzz054. PMID 30921466